CLINICAL TRIAL: NCT00699426
Title: The Effect of Nexium and Cardi-04 Yoghurt on Insulin Secretion and Effect and Cardi Vascular Risk Factors Associated With the Insulin Syndrome in Patients With Type 2 Diabetes - a Randomized Double-blind, Prospective, Placebo Controlled 2 x 2 Factorial Design 3 Month's Study.
Brief Title: The Effect of Nexium and Probiotics on Insulin Secretion and Cardiovascular Risk Factors in Patients With Type 2 Diabetes
Acronym: Nexium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lise Tarnow (Other)
Collaborators: Novo Nordisk A/S (Industry); Chr Hansen A/S (Unknown); Statens Serum Institut (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Lise Tarnow, professor, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT: 2007-00405237
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Esomeprazole; Yogurt; Placebo Effect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nexium + Yoghurt (Active Comparator)
  Interventions: Drug: nexium
- Nexium + Placebo (Placebo Comparator)
  Interventions: Drug: nexium
- Placebo+ Yoghurt (Placebo Comparator)
  Interventions: Dietary Supplement: Yoghurt
- placebo+placebo (Placebo Comparator)
  Interventions: Drug: placebo+placebo

INTERVENTIONS:
Drug: nexium — 40 mg once daily is tested together with Yoghurt
  Arms: Nexium + Yoghurt
Drug: nexium — nexium and placebo are tested
  Arms: Nexium + Placebo
Dietary Supplement: Yoghurt — Yoghurt
  Arms: Placebo+ Yoghurt
Drug: placebo+placebo — placebo and placebo are tested.
  Arms: placebo+placebo

SUMMARY:
To test the effect of Nexium and probiotics on insulin secretion and cardiovascular risk factors on type 2 diabetic patients.

Study Hypothesis:

1. Nexium causes an increased gastrin secretion that increases the insulin secretion and thereby a reduction of HbA1c
2. Probiotics changes the gut flora and bloodpressure
3. Probiotics causes a change in inflammation and thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (WHO criteria) treated with metformin and/or sulfonylureas or diet
* Males and females between 40 and 70 years
* HbA1c between 6,0-10,0
* Diabetes duration > 1 year

Exclusion Criteria:

* Kidney disease (s-creatinine above the upper limit of normal range).
* Liver disease (ALAT increase > 3 times the upper limit of the normal range of ALAT).
* Macroalbuminuria (urinary albumin excretion of > 300 mg/day).
* Heart failure(NYHA class lll or lV)
* Severe neuropathy (symptoms + vibration perception threshold > 50 measured by biothesiometer.)
* Neutropenia (neutrophil count<2.0x10/l) or anemia (hemoglobin<8mM for men or <7mM for women.
* Alcohol abuse
* Drug abuse
* Severe organic or metabolic diseases including cancer
* C-peptide< 0,3 pmol/l
* Medicine interaction
* Treatment with insulin
* PPI or other medications for ulcus diseases
* Treatment with warfarin or other coumarin derivations
* Pregnant or breastfeeding women
* Allergy to medication used in the study
* Participants may not participate in another clinical intervention trial

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
insulin secretion | 1 year

SECONDARY OUTCOMES:
blood pressure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Allan A. Vaag, MD, DMSc, Principal Investigator — Steno Diabetes Center Copenhagen

REFERENCES:
- [Derived] Hove KD, Brons C, Faerch K, Lund SS, Petersen JS, Karlsen AE, Rossing P, Rehfeld JF, Vaag A. Effects of 12 weeks' treatment with a proton pump inhibitor on insulin secretion, glucose metabolism and markers of cardiovascular risk in patients with type 2 diabetes: a randomised double-blind prospective placebo-controlled study. Diabetologia. 2013 Jan;56(1):22-30. doi: 10.1007/s00125-012-2714-y. Epub 2012 Sep 26. PMID 23011351